CLINICAL TRIAL: NCT04173130
Title: Étude Monocentrique de faisabilité d'un Nouveau Dispositif Pour le Traitement de la Fissure Anale Par Toxine Botulique (FR) Monocentric Feasibility Study for a New Medical Device for the Treatment of Anal Fissure With Botulinum Toxin (EN)
Brief Title: Monocentric Feasibility Study for a New Medical Device for the Treatment of Anal Fissure With Botulinum Toxin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dieter Hahnloser (Other)
Responsible Party: Sponsor-Investigator, Dieter Hahnloser, Professor, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: DIT_Anuscope_2019
Record Dates: First submitted 2019-11-14; First posted 2019-11-21 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Anal Fissure
MeSH Terms: conditions — Fissure in Ano | interventions — Needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injection of botulinum toxin with investigational device (Experimental)
  Interventions: Device: Anuscope with needles

INTERVENTIONS:
Device: Anuscope with needles — Injection of botulinum toxin into the anal sphincter with the investigational device (anuscope with needles).

SUMMARY:
Monocentric feasibility study for a new device for the treatment of anal fissure with botulinum toxin.

DETAILED DESCRIPTION:
Anal fissure is a common anal disease. This is a longitudinal tear in the distal part of the anal canal. The fissure provokes a spasm of the internal anal sphincter and as such pain and eventually bleeding.

There are currently 3 different treatments. All available treatments tend to relax the anal sphincter, which reduces pain and promotes fissure healing.

The first treatment consists in the local application of cream into the anal canal.

The second option is the injection of botulinum toxin into the internal or external anal sphincter. Finally the third option is a surgical intervention, most frequently a lateral sphincterotomy.

Although the usefulness of botulinum toxin to treat anal fissure has been demonstrated, the results vary. This is most likely largely due to the fact that there is no standardized way to inject botulinum toxin and that there is a significant learning curve. In addition, the gesture is not without risk for the operator.

The objective of the study is to assess the feasibility of injecting botulinum toxin into the anal canal with a new medical device for patients with anal fissure.

The trial is a mono-centric pilot study conducted on 4 patients. The study is open, prospective and all patients will be treated with the botulinum toxin injected using the new medical device.

The device (single-use) under investigation and the botulinum toxin will be made available free of charge to the patient.

ELIGIBILITY:
Inclusion Criteria:

* adult patients suffering from anal fissures for a minimum of 6 weeks.
* informed consent signed

Exclusion Criteria:

* Contraindication to the use of botulinum toxin or any known allergies
* Pregnant or breastfeeding women
* Immune deficiency, immunosuppression
* Anticoagulant treatment
* Previous pelvic radiotherapy
* Acute anal inflammation (eg.proctitis)
* Internal hemorrhoids of grade 2 or higher
* Anal fissure that did not respond to a previous treatment by botulinum toxin
* History of lateral sphincterotomy
* Cardiopulmonary disease leading to reduced function of the Cardiopulmonary system

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Feasibility of the injection of the botulin toxin with the device under investigation | This outcome will be assessed right after the use of the device under investigation, at day 1 (day of the intervention).
  The operator shall answer by yes or no. If yes, the procedure is further assessed (see outcome 2)

SECONDARY OUTCOMES:
Assessment of the procedure by the operator | This outcome will be assessed right after the use of the device under investigation, at day 1 (day of the intervention).
  The operator will assess the procedure by answering the following questions:
  How was the introduction of the anuscope ? easy-neither easy nor difficult-difficult.
  How was the positioning of the anuscope? easy-neither easy nor difficult-difficult.
  How was the deployment of the needles? easy-neither easy nor difficult-difficult.
  How was the injection of the toxin? easy-neither easy nor difficult-difficult. How was the needles retraction? easy-neither easy nor difficult-difficult.
Assessment of the patient's tolerance: visual analogic scale (VAS) | This outcome will be assessed right after the use of the device under investigation, at day 1 (day of the intervention).
  Patient assessment using a visual analogic scale (0 to 10, 0 not tolerated at all, 10 well tolerated)
Assessment of the relaxation of the internal anal sphincter | day 1, day +7, day +56
  Measurement of the relaxation using MAPLe
Assessment of the incontinence | day 1, day +7, day +56
  Score of Vaizey (0 minimum score, perfect continence; 24 = maximum score, totally incontinent)
Assessment of the healing rate | day 1, day +56
  Assessment according to the Lindsey criteria
Safety of the procedure by assessing adverse events, device deficiencies and identifying new risks | day 1, day +7, day +56
  Safety of the procedure by assessing adverse events (description of adverse events, number of participants), device deficiencies (description of the deficiency) and identifying new risks

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hahnloser, Prof., Principal Investigator — Lausanne Universitaire Hospital (CHUV)
Locations (1):
- Lausanne Universitary Hospital (CHUV), Lausanne, Canton of Vaud, Switzerland